CLINICAL TRIAL: NCT02333370
Title: A Phase Ib Dose Escalation Study of the Combination of LEE011 With Letrozole and Dose Expansion of LEE011 With Hormonal Therapy for the Treatment of Pre-(With Goserelin) and Postmenopausal Women With Hormone Receptor Positive, HER2-negative, Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011A2115C
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Hormone Receptor Positive, HER2-negative, Advanced Breast Cancer
Keywords: Advanced breast cancer; Hormone receptor positive; HER2-negative; LEE011,; Letrozole; Tamoxifen; Fulvestrant; Postmenopausal Asian women; Pre and Postmenopausal Japanese women
MeSH Terms: interventions — ribociclib; Letrozole; Tamoxifen; Fulvestrant; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LEE011 +Letrozole (Experimental): LEE011 - 3 weeks on 1 week off Letrozole 2.5mg - Once daily
  Interventions: Drug: LEE011; Drug: Letrozole
- LEE011 + Tamoxifen (Experimental): LEE011 - 3 weeks on 1 week off Tamoxifen 20mg - Once daily
  Interventions: Drug: Tamoxifen; Drug: goserelin
- LEE011 + Fulvestrant (Experimental): LEE011 - 3 weeks on 1 week off Fulvestrant 500 mg - Dosed every 28 days (Day 1 for each cycle) with 1 additional dose on Day 15 of Cycle 1
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: LEE011 — LEE011 as 50 mg and 200 mg hard gelatin oral capsules as individual patient supply packaged in bottles. LEE011 will be taken QD - days 1-21 of each 28 days cycle.
  Arms: LEE011 +Letrozole
Drug: Letrozole — 25mg
  Arms: LEE011 +Letrozole
Drug: Tamoxifen — 20 mg
  Arms: LEE011 + Tamoxifen
Drug: Fulvestrant — 500 mg
  Arms: LEE011 + Fulvestrant
Drug: goserelin
  Arms: LEE011 + Tamoxifen

SUMMARY:
The purpose of the Phase Ib is to:

1. determine the recommended dose of LEE011 in combination with a standard dose of letrozole as well as to provide additional safety and anti-tumor activity data in Asian non-Japanese patients
2. determine the recommended dose of LEE011 in combination with a standard dose of letrozole as well as to provide additional safety and activity data in Japanese patients
3. evaluate the safety and anti-tumor activity of LEE011 at the RP2D established in the dose escalation part in combination with a standard dose of letrozole, fulvestrant or tamoxifen plus goserelin in Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

* Women with advanced (locoregionally recurrent or metastatic) breast cancer not amenable to curative therapy (surgery and/or radiotherapy).
* Patient has a histologically and/or cytologically confirmed diagnosis of estrogen receptor positive and/or progesterone receptor positive breast cancer
* Patient has HER2-negative breast cancer
* Patient has adequate bone marrow and organ function

Exclusion Criteria:

* Patient who received any CDK4/6 inhibitor.
* Patient has a known hypersensitivity to any of the excipients of LEE011 or letrozole
* Patients with inflammatory breast cancer.
* Patient who received any prior systemic anti-cancer therapy (including hormonal therapy and chemotherapy) for advanced breast cancer
* Patient is currently using other anti-cancer therapy
* Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects.
* Patient who has received radiotherapy ≤ 4 weeks
* Patient has a concurrent malignancy or malignancy within 3 years
* Patient has metastases to the central nervous system (CNS).
* Patient has a known history of HIV infection

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Phase Ib Dose escalation - Frequency of dose limiting toxicities (DLTs) | first cycle (28 days)
  DLTs at each dose level associated with administration of LEE011 and letrozole
Phase Ib Dose Expansion: Number of participants with adverse events (AEs) | 18 months
  This will be defined by changes in hematology and chemistry values, vital signs and ECGs, frequency and duration of AEs, lab abnormalities and other safety parameters.
  For LEE011 and letrozole or tamoxifen or fulvestrant
Phase Ib Dose Expansion: Number of participants with serious adverse events (SAEs) | 18 months
  This will be defined by changes in hematology and chemistry values, vital signs and ECGs, frequency and duration of SAEs, lab abnormalities and other safety parameters.
  For LEE011 and letrozole or tamoxifen or fulvestrant

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) - Phase Ib dose escalation | 18 months
  This will be defined by changes in hematology and chemistry values, vital signs and ECGs, frequency and duration of AEs, lab abnormalities and other safety parameters.
  For LEE011 and letrozole or tamoxifen or fulvestrant
Number of participants with serious adverse events (SAEs) - Phase Ib dose escalation | 18 months
  This will be defined by changes in hematology and chemistry values, vital signs and ECGs, frequency and duration of SAEs, lab abnormalities and other safety parameters.
  For LEE011 and letrozole or tamoxifen or fulvestrant
Overall Response Rate (ORR) - Phase Ib dose expansion | 18 months
  Anti-tumor activity for LEE011 and letrozole or tamoxifen or fulvestrant
Clinical Benefit Rate (CBR) - Phase Ib dose expansion | 18 months
  Anti-tumor activity for LEE011 and letrozole or tamoxifen or fulvestrant
Composite Plasma pharmacokinetics (PK) parameters of LEE011 (and relevant metabolites) and letrozole - Phase Ib | C1D1, C1D2, C1D8, C1D15, C1D21, C1D22, C2D15, C3D15
  As assessed by PK parameters such as Cmax, Tmax, AUC0-24hours, accumulation ratio and Ctrough for LEE011 (and relevant metabolites) and letrozole, tamoxifen and fulvestrant
Progression Free Survival (PFS) as per RECIST v1.1- phase Ib dose expansion | 18 months
  Anti-tumor activity for LEE011 and letrozole or tamoxifen or fulvestrant
Overall Survival (OS) - Phase Ib dose expansion | 18 months
  Anti-tumor activity for LEE011 and letrozole or tamoxifen or fulvestrant
Disease Control Rate (DCR) - Phase Ib dose expansion | 18 months
  Anti-tumor activity for LEE011 and letrozole or tamoxifen or fulvestrant
Duration of Response (DOR) - Phase Ib dose expansion | 18 months
  Anti-tumor activity for LEE011 and letrozole or tamoxifen or fulvestrant

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- Novartis Investigative Site, Hong Kong, Hong Kong
- Japan (12):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Hidaka, Saitama
  - Novartis Investigative Site, Kitaadachi-gun, Saitama
  - Novartis Investigative Site, Sunto Gun, Shizuoka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Koto Ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- Novartis Investigative Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiu J, Su F, Joshi M, Masuda N, Ishikawa T, Aruga T, Zarate JP, Babbar N, Balbin OA, Yap YS. Potential value of ctDNA monitoring in metastatic HR + /HER2 - breast cancer: longitudinal ctDNA analysis in the phase Ib MONALEESASIA trial. BMC Med. 2023 Aug 15;21(1):306. doi: 10.1186/s12916-023-03017-z. PMID 37580773
- [Derived] Yap YS, Chiu J, Ito Y, Ishikawa T, Aruga T, Kim SJ, Toyama T, Saeki T, Saito M, Gounaris I, Su F, Ji Y, Han Y, Gazdoiu M, Masuda N. Ribociclib, a CDK 4/6 inhibitor, plus endocrine therapy in Asian women with advanced breast cancer. Cancer Sci. 2020 Sep;111(9):3313-3326. doi: 10.1111/cas.14554. Epub 2020 Jul 28. PMID 32619077
- See also: Related Info — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18058